CLINICAL TRIAL: NCT05322330
Title: Clinical Study of the Efficacy and Safety of XPO-1 Inhibitors in Combination With CAR-T Cells in Relapsed Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Clinical Study of XPO-1 Inhibitors Plus CAR-T Cells in Relapsed Refractory B-cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: West China Hospital (Other); The General Hospital of Western Theater Command (Other); The Affiliated People's Hospital of Ningbo University Ningbo Yinzhou People's Hospital Community (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Yixing People's Hospital (Other); Affiliated Hospital of Jiangnan University (Other); Wuxi No. 2 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/R B-NHL 01
Record Dates: First submitted 2022-03-21; First posted 2022-04-11 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Keywords: XPO-1 Inhibitor; CAR-T Cells; Relapsed Refractory B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — selinexor; Influenza Vaccines; fludarabine; Cyclophosphamide; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XPO-1 Inhibitor+CAR-T Cells (Experimental): XPO-1 Inhibitor plus CAR-T Cells
  Interventions: Drug: Selinexor; Drug: Flu; Drug: CTX; Drug: CAR-T

INTERVENTIONS:
Drug: Selinexor — 40-60mg QW,w-3～d-3,PO
  Other Names: XPO-1 Inhibitor
Drug: Flu — 25-30 mg/m2，d-5 ～d-3，qd，ivgtt
  Other Names: Fludarabine
Drug: CTX — 250-500 mg/m2，d-5 ～d-3，qd，ivgtt
  Other Names: Cyclophosphamide
Drug: CAR-T — 2-5×10^6 CAR-T/kg，ivgtt。
  Other Names: Chimeric antigen receptor-modified T (CAR-T) cell therapy

SUMMARY:
Aim of this study will evaluate the Efficacy and Safety of XPO-1 inhibitors in combination with CAR-T cells in relapsed refractory B-cell non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
B-cell non-Hodgkin's lymphoma (B-NHL) is the most common hematological malignancy originating from lymphohematopoietic tissue. Lymphoma is now one of the most rapidly growing malignancies worldwide, with approximately 350,000 new cases and over 200,000 deaths worldwide each year.With the use of rituximab in combination with standard chemotherapy regimens, progression-free survival (PFS) and overall survival (OS) in B-NHL have improved significantly, yet primary resistance or relapse progression still occurs in 40%-50% of B-NHL patients.The most widely used CAR-T therapy for R/R B-NHL in clinical practice is CAR-T therapy targeting CD19, which has a complete remission rate (CR) of 40%-53% and an overall remission rate (ORR) of 52%-82%.XPO1 inhibitors are potential drugs to enhance the anti-lymphoma effect of CD19 CAR-T cells, this study will evaluate the efficacy and safety of XPO-1 inhibitors in combination with CAR-T cells in relapsed refractory B-cell non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pathological immunohistochemistry or flow cytometry confirmed that R/ R B-cell Non-Hodgkin's Lymphoma with measurable (diameter greater than 1.5cm) lesions meets any of the following conditions: 1> After 4 courses of standard first-line therapy or 2 courses of more than two-line therapy, the lesions were reduced by <50%; 2> R/ R B-cell Non-Hodgkin's Lymphoma with disease progression after first-line or induction therapy; 3> After hematopoietic stem cell transplantation, new lesions appear or the size of previously affected lesions increased by more than 50%.
3. Previously treated with 2 or more lines of therapy.
4. ECOG≤2#.
5. The main organ functions need to meet the following conditions:LVEF≥50%;CR≤132 umol/l or CCr≥60 ml/min; ALT and AST≤2.5 times normal range#TB≤2 times ULN#Lung function≤Level 1; dyspnea(CTCAE v5.0),and blood oxygen saturation without oxygen absorption> 90%.
6. Pass the T-cell amplification test.
7. Voluntary tissue puncture/biopsy for tumor tissue retrieval before and after treatment.
8. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up one year period of the study.
9. Estimated survival time ≥3 months.
10. Voluntary signing of informed consent and good compliance.

Exclusion Criteria:

1. Have used immunosuppressants or hormones within 2 weeks prior to signing informed consent, or plan to have to use immunosuppressants or high-dose hormones (e.g. prednisone >15mg) after signing informed consent, specifically systemic treatment, excluding treatment with topical or inhaled corticosteroids.
2. The presence of bacterial, fungal, viral, mycoplasma or other types of infection that, in the judgment of the investigator, are difficult to control.
3. Active hepatitis B or active hepatitis C.
4. HIV infection.
5. Active acute or chronic graft-versus-host disease (GVHD) at the time of signing the informed consent form.
6. Participated in an investigational clinical trial of any other drug within 30 days prior to signing the informed consent form.
7. Received CAR-T cell therapy within 3 months prior to signing the informed consent form.
8. Received an allogeneic hematopoietic stem cell transplant within 6 months prior to signing the informed consent form.
9. Presence of contraindications to XPO-1 inhibitor.
10. Prior malignancy (other than Relapsed Refractory B-cell Non-Hodgkin's Lymphoma), except for cured malignant tumors with no active lesions for 3 years;Adequate treatment of inactive lesions in non-melanoma skin cancer,malignant tonsilloma or carcinoma in situ.
11. Pregnant or breasting-feeding women.
12. Conditions deemed by the researcher to be inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 12 months
  To measure the duration of response to XPO-1 Inhibitor Plus CAR-T Cells over a follow-up period of 12 months
Duration of Response(DOR) Duration of Response(DOR) | up to 12 months
  Duration of overall response will be assessed from the first XPO-1 Inhibitor Plus CAR-T cells given to progression,death or last follow-up.
Adverse events profile | up to 12 months
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated.

SECONDARY OUTCOMES:
Complete Response Rate | up to 12 months
  Number of patients who achieved complete response after treatment by XPO-1 Inhibitor plus CAR-T cells.
Progression-free Survival | up to 12 months
  To measure the duration of response to XPO-1 Inhibitor plus CAR-T cells over a follow-up period of 12 months.
Overall Survival | up to 12 months
  OS will be assessed from the first XPO-1 Inhibitor plus CAR-T cells given to death or last follow-up.
Peak Plasma Concentration | Measured from start of treatment until 28 days after last dose
  the peak amplification of CART in peripheral blood.
Time to Peak Amplification | Measured from start of treatment until 28 days after last dose
  The time to peak amplification of CART in peripheral blood.
AUC0-28 | Measured from start of treatment until 28 days after last dose
  The area under the curve (AUC0-28) obtained by plotting the number of CAR-T cells in serum against the visit time from 0 to 28 days after reinfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China